CLINICAL TRIAL: NCT02759458
Title: Evaluation of the Healicoil Suture Anchor for Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Carla Edwards, Clinical Research Manger, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12062003
Record Dates: First submitted 2016-04-21; First posted 2016-05-03 (Estimated); Results first posted 2022-09-26 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Rotator Cuff Tear Repair Anchors

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Healicoil (Experimental): Patients that met the inclusion criteria who were randomly selected to receive the Healicoil anchor for their rotator cuff repair.
  Interventions: Device: Smith & Nephew Healicoil Anchor
- Twinfix (Active Comparator): Patients that met the inclusion criteria who were randomly selected to not receive the Healicoil anchor for their rotator cuff repair.
  Interventions: Device: Smith & Nephew Twinfix Anchor

INTERVENTIONS:
Device: Smith & Nephew Healicoil Anchor
  Arms: Healicoil
Device: Smith & Nephew Twinfix Anchor
  Arms: Twinfix

SUMMARY:
The purpose of the proposed study is to evaluate a new anchor for rotator cuff repair, the Smith & Nephew Healicoil anchor. This anchor utilizes a small open-construct design to promote bone-in growth and potentially allow for the release of bone marrow factors into the repair site. In vivo ovine studies comparing the Arthrex BioComposite Corkscrew FT rotator cuff anchor to the Arthrex SwivelLock anchor have shown superior bone in-growth.

Thus, this study consists of three separate aims in order to clinically and biochemically investigate the capabilities of the Healicoil anchor and its efficacy in rotator cuff repair. One, evaluate the bone in growth of the anchor compared to a standard poly-ether ether ketone (PEEK) anchor. Two, analyze the marrow elements that are released into the repair site through the open construct. Three, compare the functional outcomes of patients with rotator cuff repairs using the Healicoil anchor compared to a traditional Twinfix PEEK anchor.

DETAILED DESCRIPTION:
A great deal of research has been devoted to determining optimal techniques for rotator cuff repair, a common orthopedic procedure. Current repair techniques involve the use of suture anchors or transosseous tunnels, with the goal of reattaching the torn tendon to the anatomic insertion of the rotator cuff. There are a multitude of different repair constructs and anchor designs available. For example, some surgeons utilize a single row of suture anchors for repair, whereas others will use two rows of anchors in a "double row" construct. A variety of anchors are also available; some are loaded with suture and require knot tying, and others can be used in a "knotless" technique. Regardless, time zero stability of the rotator cuff repair is essential, but ideal anchor or construct has yet to be determined.

Time zero stability immediately after the rotator cuff repair is important, however, contemporary research has also focused on the cascade that influences biologic healing of these rotator cuff repairs and if augmentation can improve functional results. Specifically, various authors have looked at the cytokines, growth factors and stem cells involved in the process. The question remains of what role these factors play and whether there are techniques that can facilitate their use and improve healing of rotator cuff repairs. Data exists in a animal models that does show that some of these growth factors can improve tendon healing.

Research Plan:

The proposed study will be a prospective randomized trial of 40 patients undergoing arthroscopic repair of full thickness rotator cuff tears. Patients will be randomized to one of two groups; the Healicoil anchor vs standard 5.5 PEEK anchor. Follow-up will take place at 6 weeks, 6 months, and 1 year after rotator cuff repair.

At the time of the operative procedure bone marrow aspirate from the drill hole used for the anchors will be sent for analysis. At the 6 month mark patients will get a computer tomography (CT) scan in order to determine the amount of ingrowth within the anchor. Finally, the outcome scores within the first year will be recorded. This data will result in the publication of three separate studies.

* Growth factor and stem cell analysis at the time of the operative procedure
* CT ingrowth of the Healicoil anchor at 6 months
* Clinical outcomes of patients with rotator cuff repair using the Healicoil anchor

Enrollment Process:

Patients who are determined clinically to have a full thickness rotator cuff tear and who elect to have surgery will be invited to participate in this study. Informed consent will be obtained pre-operatively in the office setting. A physical examination of both shoulders will be conducted, and all patients will complete a shoulder survey in order to determine baseline values for the Simple Shoulder Test (SST), American Shoulder and Elbow Surgeons Shoulder Score (ASES), University California, Los Angeles activity score (UCLA), and Constant scores.

Eligible patients will be randomized into one of two study groups at the time of surgery. Enrollment will continue until 20 patients are in each group. Participants in the control group will undergo rotator cuff repair utilizing 5.5mm full thread Twinfix PK anchors for tendon fixation. Those in the experimental group will undergo the same procedure, but with the use of Smith & Nephew Healicoil anchors. Participants will be blinded as to the anchor-type received.

Operative Procedure:

A standard rotator cuff repair will be completed utilizing a medial row Healicoil and a lateral row PEEK anchor. At the time of drilling for the anchors, bone marrow aspirate will be collected by turning off the water and using a large gauge biopsy needle to aspirate the contents of the drill hole. The anchors will then be placed. The aspiration process is then repeated and a smaller gauge needle will be used to aspirate within the open construct of the Healicoil anchor. All material will be sent to the laboratory of Dr. Chubinskaya for immediate analysis of:

* IGF-1
* FGF-2
* BMP-7
* BMP-2
* PDGF-CHAIN A
* PDGF-CHAIN B
* EGF
* VEGF
* Mesenchymal stem cells

Office Visits:

Following surgical rotator cuff repair, all patients will return for routine post-operative follow-up at 6 weeks, 6 months, and one year. The 6 week visit will involve a clinical exam and assessment of shoulder range of motion.

At the 6 month and 1 year visits, patients will complete the subjective and objective outcome measures and have a physical examination of both shoulders by a member of the research team. Subject participation will last approximately 30 minutes. Subjective and objective measures will include:

* Shoulder Survey - including SANE, VAS, ASES, Constant score
* Shoulder physical exam

The shoulder Survey may be collected by paper or electronically using OBERD (Rush approved repository - ORA #12042506). The shoulder Survey data which was collected up to 30 days before the time of surgery will be sued as baseline data.

CT Scanning:

At the 6 month follow up visit patients will undergo a directed CT scan of the affected humeral head only. The scan will provide 1 mm cuts through the humeral head greater tuberosity (site of anchor) only. This will limit the amount of radiation exposure to the patient and will provide the necessary data. Previous authors have shown that this technique can make the radiation exposure to the patient roughly equivalent to a standard chest xray.

These CT scans will be evaluated for the presence of bone within the confines of the anchor. One mm scanning will allow for quantitative volume analysis of the bone present.

Planned Analysis:

Descriptive statistics will be obtained for the age at time of surgery, physical examination findings, range of motion, standardized scores, bone marrow growth factor analysis, and bone in-growth as evaluated by CT scan. The statistical analysis will be conducted at a p level of < .05. Statistical tests that will be used to obtain inferential statistics of findings include paired t-tests and ANOVA.

Geoffrey S. Van Thiel, MD, MBA and Scott W. Trenhaile, MD are collaborating investigators at Rockford Orthopedics in Rockford, Illinois, Rush will subcontract with Rockford Orthopedics to enroll subjects, treat per study protocol and do follow-up visits. The bone marrow analysis of Rockford subjects will be done here at Rush. Rockford Orthopedics will use their local IRB for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is determined to have a full thickness rotator cuff tear either on pre-operative MRI scan and confirmed arthroscopically to be 1-3 cm
* Patient elects for surgical rotator cuff repair
* Written informed consent is obtained

Exclusion Criteria:

* Revision surgery
* Irreparable rotator cuff tear
* Diabetes
* Workers Compensation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01-15 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Healicoil: Patients that met the inclusion criteria who were randomly selected to receive the Healicoil anchor for their rotator cuff repair.
  Smith & Nephew Healicoil Anchor
- Twinfix: Patients that met the inclusion criteria who were randomly selected to not receive the Healicoil anchor for their rotator cuff repair.
  Smith & Nephew Twinfix Anchor
Period: Overall Study
Arm/Group | Healicoil | Twinfix
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healicoil | Twinfix | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 45 [18 to 65] | 47 [18 to 65] | 46 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder and Elbow Surgeons( ASES)-Shoulder Form
Description: This is a survey that assess the subject's current functionality and ability to complete daily tasks.
  The ASES score can be viewed as a single 100-point scale that evaluates two dimensions of shoulder function: pain and performance in activities of daily living. Each of the two domains make up for 50 of the 100 points. The higher the number on the scale, the better the pain level and subject's current functionality and ability to complete daily tasks; 100 means no shoulder pain and perfect functionality and ability to complete daily tasks.
Time Frame: 12-month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Healicoil | Twinfix
Number analyzed (Participants) | 20 | 20
score on a scale | 30 [25 to 35] | 30 [25 to 35]

2. Primary Outcome: Single Assessment Numeric Evaluation (SANE) Form
Description: This is a single question survey that asks how the patient's shoulder is feeling.
  The Single Assessment Numeric Evaluation (SANE) is a patient rating from 0-100. Patients rate their current illness score in relation to their pre-injury baseline.
  The higher the number on the scale, the better the patient's shoulder is feeling compared to their pre-injury baseline. 100 means the patient's shoulder feels in perfect health compared with pre-injury baseline.
Time Frame: 12-month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Healicoil | Twinfix
Number analyzed (Participants) | 20 | 20
score on a scale | 50 [45 to 55] | 48 [45 to 55]

ADVERSE EVENTS:
Arm/Group | Healicoil | Twinfix
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No